CLINICAL TRIAL: NCT01033747
Title: A 5-year Open Label, Non-comparative Extension to a Randomized, Open-label, Phase IIa Study to Evaluate Safety, Tolerability and the Effects on Liver Iron Concentration of Repeated Doses of 10 and 20 mg/kg/Day of Deferasirox in Comparison With 40 mg/kg/Day Deferoxamine in Patients With Transfusion-dependent Iron Overload
Brief Title: Safety and Efficacy of Deferasirox in Patients With Transfusion Dependent Iron Overload - a Non-comparative Extension Study
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CICL670A0105E2
Record Dates: First submitted 2009-10-16; First posted 2009-12-16 (Estimated); Results first posted 2011-08-11 (Estimated); Last update posted 2011-08-11 (Estimated); Status verified 2011-07

CONDITIONS: Liver Iron Overload
Keywords: iron overload; iron chelation therapy; B-thalassemia
MeSH Terms: conditions — Iron Overload; beta-Thalassemia | interventions — Deferasirox

ARMS (2):
- Deferasirox (Experimental): Deferasirox group consists of all participants who were initially randomized to 10 and 20 mg/kg/day deferasirox orally daily in the main study and remained on the same treatment during the comparative prolongation study (NCT00379483) and at the beginning of the 5-year non-comparative study
  Interventions: Drug: Deferasirox
- Deferasirox Crossover (Experimental): Deferasirox Crossover group consists of participants who were initially randomized to 40 mg/kg/day deferoxamine (DFO)subcutaneously in the main study and comparative prolongation study and crossed over to 5mg/kg/day to 30 mg/kg/day deferasirox orally daily at the beginning of the 5-year non-comparative extension study
  Interventions: Drug: Deferasirox

INTERVENTIONS:
Drug: Deferasirox — 10 mg/kg or 30 mg/kg orally daily
  Arms: Deferasirox
Drug: Deferasirox — 5 mg/kg or 30 mg/kg orally daily
  Arms: Deferasirox Crossover

SUMMARY:
The purpose of this study is to assess the safety and the effects on liver iron of Deferasirox when given for a long treatment period in patients with transfusion dependent iron overload.

ELIGIBILITY:
Inclusion Criteria:

* Patients Currently participating in the 9-month comparative prolongation of extension phase of the original study.
* Patients currently participating in the food-effect sub-study, according to amendment 3.
* Ability to provide written informed consent prior to participation in this non-comparative extension study.
* Female patients sexually active must use double-barrier contraception, oral contraceptive plus barrier contraceptive, or must have undergone clinically documented total hysterectomy and/or ovariectomy, or tubal ligation.
* Body weight of at least 35 kg.

Exclusion Criteria:

* Pregnant or breastfeeding patients.
* History of non-compliance to medical regimens and patients who are considered potentially unreliable.
* Proteinuria > 300 mg/L second void morning urine.
* Patients with serum creatinine above the upper limit normal.

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2003-02; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (4):
- Italy (4):
  - Novartis Investigative Site, Cagliari
  - Novartis Investigative Site, Genova
  - Novartis Investigative Site, Milan
  - Novartis Investigative Site, Torino

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This 5 year extension study includes participants treated in one or more studies: a 1 year main study to evaluate the safety,tolerability and the effects of 2 doses of deferasirox on liver iron content in comparison to standard chelation therapy with DFO, a 3 week food effect sub-study and a 12-21 month prolongation phase(NCT00379483).
Groups:
- Deferasirox: Deferasirox group consists of all participants who were initially randomized to 10 mg/kg or 20 mg/kg deferasirox orally daily in the main study and remained on deferasirox treatment during the comparative prolongation study (NCT00379483) and at the beginning of the 5-year non-comparative extension study
- Deferasirox Crossover: Deferasirox Crossover group consists of participants who were initially randomized to 40 mg/kg/day deferoxamine (DFO) subcutaneously in the main study and comparative prolongation study and crossed over to 5 mg to 30 mg/kg/day deferasirox orally daily at the beginning of the 5-year non-comparative extension study
Period: Overall Study
Arm/Group | Deferasirox | Deferasirox Crossover
Started | 51 | 19
Completed | 14 | 4
Not Completed | 37 | 15
Not completed — Adverse Event | 9 | 4
Not completed — Abnormal Laboratory Value | 1 | 0
Not completed — Abnormal test procedure | 0 | 1
Not completed — Unsatisfactory therapeutic effect | 14 | 4
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 9 | 6
Not completed — Stopped at end of prolongation visit 1 | 1 | 0
Not completed — Stopped at end of Extension 1 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Deferasirox | Deferasirox Crossover | Total
Number analyzed (Participants) | 51 | 19 | 70
Age Continuous [Mean (Standard Deviation); unit: years] | 24.7 (5.43) | 23.8 (3.76) | 24.5 (5.02)
Age, Customized [Number; unit: participants]
  16 to 49 | 50 | 19 | 69
  50 to 65 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 10 | 45
  Male | 16 | 9 | 25
Region of Enrollment [Number; unit: participants]
  Italy | 51 | 19 | 70

OUTCOME MEASURES:

1. Primary Outcome: The Relative Change From Baseline in Liver Iron Content (LIC) After Prolonged Use of Deferasirox
Description: The mean percentage change in liver iron content (LIC) as assessed by superconducting quantum interference device (SQUID) was evaluated by comparing the LIC at the start of Deferasirox treatment to the LIC at the end of the 5 year extension study for participants who were treated with Deferasirox for more than 3.5 years. LIC is expressed in milligrams of iron per gram of liver dry weight (mgFe/g dw). Relative change = 1- (Change in LIC from Baseline/Baseline level) x 100.
Time Frame: Baseline to 7 Years
Population: All participants in the full analysis set treated with deferasirox for more than 3.5 years.
Measure: Mean (Full Range); unit: Percent change
Arm/Group | Deferasirox | Deferasirox Crossover
Number analyzed (Participants) | 36 | 8
Percent change | -21.9 (47.11) [-97.1 to 124.6] | -23.1 (33.38) [-62.2 to 18.8]

2. Secondary Outcome: Relative Change in Serum Ferritin From Baseline to 3.5 Years
Description: The mean percentage change in serum ferritin was evaluated by comparing the serum ferritin level at the start of Deferasirox treatment to the serum ferritin level collected 18 months following the start of the extension study. Serum ferritin is measured in micrograms per Liter. Relative Change = 1- (Change in ferritin level from Baseline/Baseline level) x 100.
Time Frame: Baseline to 3.5 years
Population: All participants comprised of the full analysis set were evaluated for the change in serum ferritin.
Measure: Mean (Full Range); unit: Percent change
Arm/Group | Deferasirox | Deferasirox Crossover
Number analyzed (Participants) | 51 | 19
Percent change | 32.4 [-68.8 to 152.7] | 33.2 [-10.0 to 99.8]

ADVERSE EVENTS:
Groups:
- Deferasirox: Deferasirox group consists of all participants who were initially randomized to 10 mg/kg or 20 mg/kg deferasirox orally daily in the main study and remained on the same deferasirox treatment during the comparative prolongation study(NCT00379483)and at the beginning of the 5-year non-comparative extension study
- Deferasirox Crossover: Deferasirox Crossover group consists of participants who were initially randomized to 40 mg/kg/day deferoxamine (DFO)subcutaneously in the main study and comparative prolongation study and crossed over to 5 mg/kg to 30 mg/kg deferasirox orally daily at the beginning of the 5-year non-comparative extension study.
Arm/Group | Deferasirox | Deferasirox Crossover
Serious Adverse Events (participants affected / at risk) | 18/51 | 2/19
Other Adverse Events (participants affected / at risk) | 50/51 | 19/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Deferasirox (N=51) | Deferasirox Crossover (N=19)
Extramedullary haemopoiesis (Blood and lymphatic system disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Chest pain (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Bacterial infection (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Bronchopneumonia (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1
Nasal abscess (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Injury (Injury, poisoning and procedural complications) | 1 | 0
Neck injury (Injury, poisoning and procedural complications) | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0
Tendon injury (Injury, poisoning and procedural complications) | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0
Metabolic disorder (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Tendon disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Monoparesis (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Renal colic (Renal and urinary disorders) | 3 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal turbinate hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cholecystectomy (Surgical and medical procedures) | 1 | 0
Splenectomy (Surgical and medical procedures) | 1 | 0
Surgery (Surgical and medical procedures) | 1 | 0
Thrombophlebitis (Vascular disorders) | 2 | 0
Venous thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Deferasirox (N=51) | Deferasirox Crossover (N=19)
Lymphadenopathy (Blood and lymphatic system disorders) | 3 | 0
Cardiac failure (Cardiac disorders) | 2 | 1
Palpitations (Cardiac disorders) | 7 | 1
Tachycardia (Cardiac disorders) | 6 | 5
Ear pain (Ear and labyrinth disorders) | 5 | 2
Vertigo (Ear and labyrinth disorders) | 9 | 4
Hypogonadism (Endocrine disorders) | 5 | 0
Chalazion (Eye disorders) | 3 | 0
Conjunctivitis (Eye disorders) | 3 | 0
Conjunctivitis allergic (Eye disorders) | 5 | 2
Eyelid oedema (Eye disorders) | 0 | 1
Scotoma (Eye disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 3
Abdominal pain (Gastrointestinal disorders) | 24 | 5
Abdominal pain upper (Gastrointestinal disorders) | 22 | 6
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 3 | 4
Diarrhoea (Gastrointestinal disorders) | 20 | 8
Dyspepsia (Gastrointestinal disorders) | 9 | 2
Enteritis (Gastrointestinal disorders) | 8 | 3
Gastritis (Gastrointestinal disorders) | 6 | 2
Nausea (Gastrointestinal disorders) | 19 | 4
Rectal prolapse (Gastrointestinal disorders) | 0 | 1
Toothache (Gastrointestinal disorders) | 8 | 1
Vomiting (Gastrointestinal disorders) | 16 | 1
Asthenia (General disorders) | 20 | 4
Chest discomfort (General disorders) | 1 | 1
Chest pain (General disorders) | 4 | 2
Gravitational oedema (General disorders) | 0 | 1
Influenza like illness (General disorders) | 9 | 1
Oedema peripheral (General disorders) | 10 | 0
Pyrexia (General disorders) | 31 | 9
Bronchitis (Infections and infestations) | 12 | 1
Cystitis (Infections and infestations) | 4 | 2
Dysentery (Infections and infestations) | 1 | 1
Ear infection (Infections and infestations) | 3 | 2
Fungal skin infection (Infections and infestations) | 2 | 2
Gastroenteritis (Infections and infestations) | 9 | 2
Hordeolum (Infections and infestations) | 3 | 0
Influenza (Infections and infestations) | 25 | 7
Localised infection (Infections and infestations) | 1 | 1
Nasopharyngitis (Infections and infestations) | 17 | 5
Oral herpes (Infections and infestations) | 3 | 0
Paronychia (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 34 | 6
Pharyngotonsillitis (Infections and infestations) | 2 | 2
Rhinitis (Infections and infestations) | 29 | 7
Sinusitis (Infections and infestations) | 6 | 1
Tonsillitis (Infections and infestations) | 7 | 3
Tooth abscess (Infections and infestations) | 9 | 1
Tooth infection (Infections and infestations) | 0 | 1
Tracheitis (Infections and infestations) | 6 | 1
Urinary tract infection (Infections and infestations) | 7 | 3
Vaginal infection (Infections and infestations) | 6 | 0
Vulvovaginal candidiasis (Infections and infestations) | 0 | 1
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 1
Wound infection (Infections and infestations) | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 2 | 1
Muscle strain (Injury, poisoning and procedural complications) | 1 | 1
Neck injury (Injury, poisoning and procedural complications) | 0 | 2
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 1
Skeletal injury (Injury, poisoning and procedural complications) | 3 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 1
Transfusion reaction (Injury, poisoning and procedural complications) | 4 | 1
Beta 2 microglobulin increased (Investigations) | 6 | 0
Beta 2 microglobulin urine increased (Investigations) | 4 | 0
Blood folate decreased (Investigations) | 2 | 1
Blood phosphorus decreased (Investigations) | 0 | 1
Blood thyroid stimulating hormone increased (Investigations) | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 3 | 0
Transaminases increased (Investigations) | 4 | 1
Vitamin C decreased (Investigations) | 8 | 1
Vitamin E decreased (Investigations) | 4 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1
Zinc deficiency (Metabolism and nutrition disorders) | 4 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 16 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 29 | 9
Bone pain (Musculoskeletal and connective tissue disorders) | 8 | 3
Flank pain (Musculoskeletal and connective tissue disorders) | 4 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 7 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 7 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 3 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10 | 2
Torticollis (Musculoskeletal and connective tissue disorders) | 2 | 1
Dizziness (Nervous system disorders) | 5 | 1
Headache (Nervous system disorders) | 29 | 9
Hypoaesthesia (Nervous system disorders) | 1 | 1
Paraesthesia (Nervous system disorders) | 2 | 3
Presyncope (Nervous system disorders) | 8 | 1
Sciatica (Nervous system disorders) | 5 | 2
Anxiety (Psychiatric disorders) | 4 | 0
Depression (Psychiatric disorders) | 4 | 0
Insomnia (Psychiatric disorders) | 4 | 1
Dysuria (Renal and urinary disorders) | 7 | 1
Glycosuria (Renal and urinary disorders) | 1 | 1
Micturition disorder (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 5 | 0
Nephropathy toxic (Renal and urinary disorders) | 1 | 2
Nocturia (Renal and urinary disorders) | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 2
Proteinuria (Renal and urinary disorders) | 0 | 1
Renal colic (Renal and urinary disorders) | 7 | 1
Renal tubular disorder (Renal and urinary disorders) | 0 | 1
Strangury (Renal and urinary disorders) | 2 | 1
Amenorrhoea (Reproductive system and breast disorders) | 4 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 3 | 1
Genital discharge (Reproductive system and breast disorders) | 1 | 1
Genital haemorrhage (Reproductive system and breast disorders) | 0 | 2
Pruritus genital (Reproductive system and breast disorders) | 0 | 1
Vulvovaginal pruritus (Reproductive system and breast disorders) | 2 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 36 | 7
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 23 | 7
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Erythema (Skin and subcutaneous tissue disorders) | 3 | 0
Koilonychia (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 2
Rash (Skin and subcutaneous tissue disorders) | 2 | 3
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 3 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 4 | 0
Tooth extraction (Surgical and medical procedures) | 0 | 1
Hypotension (Vascular disorders) | 5 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.